CLINICAL TRIAL: NCT01384721
Title: Computed Tomography Coronary Angiography Prognostic Registry for Coronary Artery Disease - CTCA-PRORECAD
Brief Title: Computed Tomography Coronary Angiography (CTCA) Prognostic Registry for Coronary Artery Disease
Acronym: PRORECAD
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Collaborators: Società Italiana di Radiologia Medica (Other)
Responsible Party: Principal Investigator, Filippo Cademartiri, Associate Professor, Azienda Ospedaliero-Universitaria di Parma
Other Study IDs: SIRM-PRORECAD
Record Dates: First submitted 2011-06-28; First posted 2011-06-29 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Coronary Artery Disease; Atherosclerosis
Keywords: Computed Tomography Coronary Angiography; Coronary Artery Disease; Prevalence Of Disease; Prognosis; Risk Stratification
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study aims at pooling a large population of patients with suspected coronary artery disease (CAD) who underwent Computed Tomography Coronary Angiography (CTCA) and who were adequately stratified in the first place. Then the investigators will be able to assess the incremental value of CTCA in the stratification of prevalence of disease (non obstructive/obstructive) and prognosis of patients with suspected CAD). The added information to current evidence is how reliable and to what extent CTCA can define the actual burden of disease and cardiovascular risk.

DETAILED DESCRIPTION:
The Project aims at pooling (retrospectively) a large population of patients with suspected coronary artery disease (CAD) who underwent Computed Tomography Coronary Angiography (CTCA) and who were adequately stratified in the first place. Then the investigators will be able to assess the incremental value of CTCA in the stratification of prevalence of disease (non obstructive/obstructive) and prognosis of patients with suspected CAD. The added information to current evidence is how reliable and to what extent CTCA can define the actual burden of disease and cardiovascular risk.

Primary objectives

* MACE/Major Adverse Cardiovascular Events (i.e. Cardiac Death, Unstable Angina requiring Hospitalization, Acute Myocardial Infarction)
* Prevalence of cardiovascular risk category shifting based on coronary plaque burden

Secondary objectives

* Coronary Revascularizations occurred after CTCA (i.e. PCI/Percutaneous Coronary Revascularization and CABG/Coronary Artery Bypass Graft)
* Prevalence of outliers (i.e. patients lying completely outside the conventional risk stratification; pts with >3 risk factors and no CAD at CTCA and pts with no risk factors and >5 coronary segments with CAD)

Institutional Database will be used as data supply. Data will be anonimyzed and pooled (i twill not be possible to detect patients' identity). For this reason the investigators will no task for patients' Informed Consent.

DESIGN The investigators will retrospectively collect data from respective Institutional databases regarding patients who underwent CTCA for suspected CAD in the last 4 years.

General Inclusion criteria Only patients with also Calcium Score

≥64-slice CT technology (or 16-slice CT technology with >4 year follow-up) Number of patients of at least 100 with complete clinical file and follow-up Minimum follow-up of 12 months Only patients with suspected Coronary Artery Disease

METHODS Study design and patient population This is an observational retrospective study (consecutive patients meeting the inclusion criteria) in patients with suspected coronary artery disease referred to our Institutions for evaluation by Computed Tomography Coronary Angiography (CTCA) starting in January 2003. Participating centers will provide data from 16-slice CTCA (minimum follow-up >4 years) or superior (i.e. 64-slice CTCA; minimum follow-up 12 months). Each center will have to provide at least 200 patients (with complete file for evaluation).

Patients are usually referred because of symptoms (chest pain, dyspnoea on exertion) and/or abnormal or equivocal stress test and/or high cardiovascular risk profile. Exclusion criteria are renal failure (creatinine clearance <60ml/min), known previous reaction to iodinated contrast medium and pregnancy, history of Myocardial Infarction, previous revascularization (PCI and/or CABG).

All the patients will be assessed by interview and by data collection from clinical database of the Institution for presence of cardiovascular risk factors and symptoms. The following risk factors will be considered: 1) Hypertension (defined as Arterial Pressure 140/80 mmHg or need for antihypertensive therapy); 2) Hypercholesterolemia (LDL Cholesterol >130 mg/dl or current treatment with lipid-lowering therapy); 3) Diabetes Mellitus (current need for antidiabetic or insulin therapy); 4) Smoking habit; 5) Obesity (Body Mass Index/BMI> 30); 6) Family history of cardiac disease. Symptoms will be classified as no symptoms, typical chest pain, atypical chest pain, dyspnoea on exertion. The pre-test cardiovascular risk of the patients will be determined by means of the Morise risk score.

Follow-up Follow-up data of all the patients were obtained by outpatient visit and/or phone contact and/or data collection from clinical database of the Institution. Minimum follow-up will be 6 months. Hospital/patients' records were screened for the occurrence of clinical events to confirm the obtained information. The clinical end-points are: 1) cardiac death, 2) non-fatal acute myocardial infarction, 3) unstable angina requiring hospitalization, 4) percutaneous or surgical revascularization. Cardiac death is defined as death caused by acute myocardial infarction or ventricular arrhythmias. Non-fatal myocardial infarction is defined based on criteria of typical chest pain, elevated cardiac enzyme levels, and typical changes on the electrocardiogram. Revascularization is defined as percutaneous coronary intervention (PCI) with stenting or coronary artery bypass surgery (CABG). The end point was the occurrence of one MACE at follow-up.

Multislice computed tomography data acquisition All examinations were performed with a 16-slice or higher CT system (Multi-vendor). First, a prospectively triggered coronary calcium CT data set was obtained using standardized CT parameters. Thereafter CTCA was performed after the administration of a bolus (60-100ml) non ionic contrast material (Multi-vendor) at flow rate of 4-6ml/s depending on patient status. All injections were performed by power injector via an antecubital vein and were followed by 50 ml of saline bolus chase at the same flow rate. A bolus tracking technique was used to determine the initiation of CT data acquisition. CTCA was performed with the best available parameters, depending on scanner type and generation. The reconstruction slice thickness and increment were 0.5-0.75mm and 0.3-0.5mm respectively. Intra-venous beta-blocker (e.g. atenolol 5-10mg) was administered to all patients with a heart rate >65 beats/min and without contraindication (known asthma or bronchospasm, systolic blood pressure <100mmHg). In addition, nitro-glycerine was administered sublingually to all patients, albeit contraindications (known significant aortic stenosis, systolic blood pressure <100mmHg). Patients with atrial fibrillation or frequent premature beats were included in the study. To obtain optimal image quality, datasets were reconstructed at least at two points of the cardiac cycle using a retrospective ECG gating algorithm (one diastolic cardiac phase usually at -350msec from the R waves and one end-systolic phase at +275msec). In the presence of motion artefacts, as in the case of cardiac arrhythmias, additional reconstructions were made at different time points of the R-R interval. At the time of the study, tube current modulation was not used. The estimated radiation dose would be 5-20mSv. Axial data sets are transferred to a remote workstation (Multi-vendor) for post-processing and subsequent evaluation.

CTCA data analysis - Coronary Artery Calcium Score The coronary artery calcium (CACS) score was assessed with the application of dedicated software (Multi-vendor). Coronary artery calcium was identified as a dense area in the coronary artery whose attenuation exceeded the threshold of 130 Hounsfield units (HU). The overall calcium score was calculated according to Agatston score algorithm for each patient.

CTCA data analysis - Coronary Artery Atherosclerotic plaque assessment All CTCA angiograms are evaluated locally by 2 experienced board certified observers. In case of disagreement, a joint reading was performed and a consensus was reached. Coronary arteries were divided into 15-16 segments according to the modified American Heart Association classification and in the case the intermediate branch was present it was added to the classification. All coronary segments were considered in the analysis. First, each segment was classified as assessable or not assessable. All assessable segments were then evaluated for the presence of any atherosclerotic plaque. Axial images and curved multiplanar reconstructions of the segmental vasculature were utilized for the assessment. Coronary plaques were defined as described previously as structures of >1mm^2 within and/or adjacent to the coronary artery lumen which are clearly distinguishable from the vessel lumen and surrounding pericardial tissue. Obstructive coronary plaques were defined as plaques resulting in ≥50% luminal narrowing; non obstructive plaques were defined as plaques that resulted in <50% luminal narrowing. Patients were classified as belonging to one of three groups based on the CTCA findings: 1) patients with normal coronary arteries, 2) patients with non obstructive coronary artery disease, and 3) patients with obstructive coronary artery disease (presence of at least one plaque ≥50%).

Statistical analysis Categorical baseline characteristics, expressed as numbers and percentages, will be compared using the chi-square test. Continuous variables, expressed as mean and standard deviation (SD), will be compared using the 2-tailed t test and analysis of variance if normally distributed or by means of the Kruskal-Wallis method if not normally distributed. A composite end-point of MACE will be used (cardiac death, non-fatal infarction, unstable angina). Cumulative event rates as a function of time were obtained by means of the Kaplan-Meier method. Event curves of MACE will be compared using the log-rank test. Cox regression analysis will be used to identify associations between clinical characteristics and CTCA variables and outcome. Univariate and multivariate analyses will be performed to identify potential predictors. In the multivariate analysis will be included only variables which were significant at univariate analysis. Hazard ratios will be calculated with 95% confidence intervals as an estimate of the risk associated with a particular variable. Statistical analyses will be performed using Excel 2007 software (Microsoft, United States), MedCalc software (version 8.0, United States), STATA software (version 10, United States), SPSS software (version 12.0, United States). p values <0.05 will be considered statistically significant.

Incremental value of CTCA above CACS will be analyzed. Sub-analysis for the pre-test cardiovascular risk stratification according to the Morise score (low-risk, intermediate risk, high risk) will be performed.

Sample size Based on our experience and data from literature the investigators estimated a sample size of 1000 patients. Considering the retrospective nature of the study, it is possible that at the end the investigators will reach a population >1000 patients which will anyway let the study continue to the expected 2 years duration.

ELIGIBILITY:
Inclusion Criteria:

* Only patients with also Calcium Score
* ≥64-slice CT technology (or 16-slice CT technology with >4 year follow-up)
* Number of patients of at least 100 with complete clinical file and follow-up
* Minimum follow-up of 12 months
* Only patients with suspected Coronary Artery Disease

Exclusion Criteria:

* renal failure (creatinine clearance <60ml/min)
* known previous reaction to iodinated contrast medium and pregnancy
* history of Myocardial Infarction
* previous revascularization (PCI and/or CABG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to CT Coronary angiography for suspected obstructive Coronary Artery Disease based on high cardiovascular risk and/or symptoms and/or test abnormalities
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-09; Primary Completion 2022-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
MACE/Major Adverse Cardiovascular Events | at least 12 months
  Cardiac Death, Unstable Angina requiring Hospitalization, Acute Myocardial Infarction
Cardiovascular risk shifting | at time 0
  Prevalence of cardiovascular risk category shifting based on coronary plaque burden

SECONDARY OUTCOMES:
Coronary Revascularizations | after more than 90 days
  Coronary Revascularizations occurred at follow-up after CTCA (i.e. PCI/Percutaneous Coronary Revascularization and CABG/Coronary Artery Bypass Graft)
Prevalence of outliers | at time 0
  Prevalence patients lying completely outside the conventional risk stratification (pts with >3 risk factors and no CAD at CTCA and pts with no risk factors and >5 coronary segments with CAD)

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Cademartiri, MD, PhD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma, Italy
Locations (11):
- Italy (11):
  - Policlinico San Donato IRCCS, Milan, MI
  - Dibimel, Department of Radiology, University of Palermo, Palermo, PA
  - Azienda Ospedaliero-Universitaria di Parma, Parma, PR
  - Department of Radiology - Area Vasta 1 - ASUR Marche, Urbino, PU
  - Cardiothoracovascular Department cardiovascular radiology Unit, University Hospital Bologna, Bologna
  - AUSL n. 1 Toscana - Ospedale di Carrara, Carrara
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - Sdn Irccs, Naples
  - San Gennaro Hospital, Naples
  - University of Rome "Sapienza", Polo Pontino, Rome
  - Università Sapienza di Roma, Rome

REFERENCES:
- [Background] Maffei E, Seitun S, Martini C, Aldrovandi A, Cervellin G, Tedeschi C, Guaricci A, Messalli G, Catalano O, Cademartiri F. Prognostic value of computed tomography coronary angiography in patients with chest pain of suspected cardiac origin. Radiol Med. 2011 Aug;116(5):690-705. doi: 10.1007/s11547-011-0647-z. Epub 2011 Mar 7. English, Polish. PMID 21424322
- [Background] Aldrovandi A, Maffei E, Seitun S, Martini C, Berti E, Grilli R, Messalli G, Weustink AC, Mollet NR, Nieman K, Ardissino D, de Feyter PJ, Krestin GP, Cademartiri F. Major adverse cardiac events and the severity of coronary atherosclerosis assessed by computed tomography coronary angiography in an outpatient population with suspected or known coronary artery disease. J Thorac Imaging. 2012 Jan;27(1):23-8. doi: 10.1097/RTI.0b013e3181f55d0d. PMID 21052023
- [Background] Maffei E, Seitun S, Martini C, Aldrovandi A, Arcadi T, Clemente A, Messalli G, Malago R, Weustink A, Mollet N, Nieman K, Ardissino D, de Feyter P, Krestin G, Cademartiri F. Prognostic value of CT coronary angiography: focus on obstructive vs. nonobstructive disease and on the presence of left main disease. Radiol Med. 2011 Feb;116(1):15-31. doi: 10.1007/s11547-010-0592-2. Epub 2010 Oct 6. English, Italian. PMID 20927651
- [Background] Aldrovandi A, Maffei E, Palumbo A, Seitun S, Martini C, Brambilla V, Zuccarelli A, Tarantini G, Weustink AC, Mollet NR, Ruffini L, Crisi G, Ardissino D, de Feyter PJ, Krestin GP, Cademartiri F. Prognostic value of computed tomography coronary angiography in patients with suspected coronary artery disease: a 24-month follow-up study. Eur Radiol. 2009 Jul;19(7):1653-60. doi: 10.1007/s00330-009-1344-3. Epub 2009 Feb 18. PMID 19224218
- [Background] Van Werkhoven JM, Cademartiri F, Seitun S, Maffei E, Palumbo A, Martini C, Tarantini G, Kroft LJ, de Roos A, Weustink AC, Jukema JW, Ardissino D, Mollet NR, Schuijf JD, Bax JJ. Diabetes: prognostic value of CT coronary angiography--comparison with a nondiabetic population. Radiology. 2010 Jul;256(1):83-92. doi: 10.1148/radiol.1090600. PMID 20574086
- [Derived] Maffei E, Midiri M, Russo V, Rengo M, Tedeschi C, Spagnolo P, Seitun S, Francone M, Guaricci AI, Carrabba N, Malago R, Cuocolo A, Arcadi T, Catalano OA, Cademartiri F. Rationale, design and methods of CTCA-PRORECAD (Computed Tomography Coronary Angiography Prognostic Registry for Coronary Artery Disease): a multicentre and multivendor registry. Radiol Med. 2013 Jun;118(4):591-607. doi: 10.1007/s11547-012-0912-9. Epub 2013 Jan 28. PMID 23358817
- See also: Website of Italian Society of Medical Radiology — http://www.sirm.org/